CLINICAL TRIAL: NCT05152966
Title: PersAFOne II(Pronounced Per-'Se-fa-nē 2); Feasibility Study of the FARAPULSE™ Cardiac Ablation System Plus in the Treatment of Persistent Atrial Fibrillation
Brief Title: Feasibility Study of the FARAPULSE™ Cardiac Ablation System Plus in the Treatment of Persistent Atrial Fibrillation(PersAFOne II)
Acronym: PersAFOne II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1335
Record Dates: First submitted 2021-11-15; First posted 2021-12-10 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- FARAPULSE™ Endocardial Cardiac Ablation (Experimental): Ablation using FARAPULSE™ Cardiac Ablation System Plus
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Ablation using the FARAPULSE™ Cardiac Ablation System Plus

SUMMARY:
The objective of this safety and feasibility study is to assess whether the endocardial creation of electrically nonconductive lesions via PEF catheter ablation applied using the FARAPULSE Cardiac Ablation System Plus is a feasible and safe treatment for PersAF and associated AFL

DETAILED DESCRIPTION:
This is a prospective, multi-center safety and feasibility study in subjects with persistent AF. Subjects will undergo percutaneous PEF ablation for pulmonary vein isolation as well as cavotricuspid isthmus interruption and other left atrial ablations at the investigator's discretion. Subjects will then be followed at 30 days, 60 ± 15 days, 6 months and 12 months for adverse events, recurrence of arrhythmia after a 90 day blanking period and other relevant outcome measures.

ELIGIBILITY:
Key Inclusion Criteria: Patients are required to meet all the following inclusion criteria to participate in this study:

* Age 18-75 Patients with documented drug-resistant symptomatic persistent AF

  1. Patient is refractory or intolerant to at least one Class I/III antiarrhythmic agent.
  2. ECG-documented first episode of persistent AF, lasting longer than 7 days but not longer than 365 days
  3. Holter within 90 days prior to the Enrollment Date demonstrating 24 hours of continuous AF 3. Patient participation requirements:

  <!-- -->

  1. Lives locally
  2. Is willing and capable of providing Informed Consent to undergo study procedures
  3. Is willing to participate in all examinations and follow-up visits and tests associated with this clinical study.

Exclusion Criteria:

Subjects will be excluded from participating in this study if they meet any one of the following exclusion criteria:

1. AF that is:

   1. Paroxysmal (longest AF episode < 7days)
   2. Longstanding (has persisted > 12 months or that does not respond to cardioversion if < 12 months)
   3. Secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible / non-cardiac causes
2. Left atrial anteroposterior diameter ≥ 5.5 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT)
3. Any of the following cardiac procedures, implants or conditions:

   1. Clinically significant arrhythmias other than AF, AFL or AT
   2. Hemodynamically significant valvular disease
   3. Prosthetic heart valve
   4. NYHA Class III or IV CHF
   5. Previous endocardial or epicardial ablation or surgery for AF
   6. Atrial or ventricular septal defect closure
   7. Atrial myxoma
   8. Left atrial appendage device or occlusion
   9. Pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices
   10. Significant or symptomatic hypotension
   11. Bradycardia or chronotropic incompetence
   12. History of pericarditis
   13. History of rheumatic fever
   14. History of congenital heart disease with any residual anatomic or conduction abnormality
4. Any of the following within 3 months prior toenrollment:

   1. Myocardial infarction
   2. Unstable angina
   3. Percutaneous coronary intervention
   4. Heart surgery (e.g. coronary artery bypass grafting, ventriculotomy, atriotomy)
   5. Heart failure hospitalization
   6. Stroke or TIA
   7. Clinically significant bleeding
   8. Pericarditis or pericardial effusion
   9. Left atrial thrombus
5. History of blood clotting or bleeding abnormalities.
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Contraindications to CT or MRI
8. Sensitivity to contrast media not controlled by premedication
9. Women of childbearing potential who are pregnant, lactating or not using birth control
10. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to

    1. Body mass index (BMI) > 40
    2. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
    3. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
    4. Renal insufficiency with an estimated creatinine clearance <30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
    5. Active malignancy or history of treated cancer within 24 months of enrollment
    6. Clinically significant gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
    7. Clinically significant infection
    8. Predicted life expectancy less than one year
11. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the protocol requirements
12. Current or anticipated enrollment in any other clinical study
13. Employment by FARAPULSE or the same hospital department or office of any investigator, or a family member of any of the preceding groups.
14. Use of amiodarone after day of index ablation procedure. Patients will cease use of amiodarone on or before the date of the index ablation procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nemocnice Na Homolce, Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FARAPULSE™ Endocardial Cardiac Ablation
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | FARAPULSE™ Endocardial Cardiac Ablation
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 20

OUTCOME MEASURES:

1. Primary Outcome: Composite Safety Endpoint;Proportion of Intent to Treat Subjects With One or More of the Specified Device or Procedure Related SAEs
Description: Proportion of Intent to Treat subjects with one or more of the specified device or procedure related SAEsEndpoint(CSE) defined as the incidence of the following early-onset serious adverse events (SAEs) which are device- or procedure-related, as adjudicated by the Clinical Events and Data Monitoring Committee (CEDMC). Atrioesophageal fistula and PV stenosis components will be assessed for occurrence at any time during follow-up.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | FARAPULSE™ Endocardial Cardiac Ablation
Number analyzed (Participants) | 20
participants | 0

2. Primary Outcome: Composite Safety Endpoint;Proportion of Intent to Treat Subjects With One or More of the Specified Device or Procedure Related SAEs
Description: Proportion of Intent to Treat subjects with one or more of the specified device or procedure related SAEsEndpoint(CSE) defined as the incidence of the following late-onset serious adverse events (SAEs) which are device- or procedure-related, as adjudicated by the Clinical Events and Data Monitoring Committee (CEDMC).
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE™ Endocardial Cardiac Ablation
Number analyzed (Participants) | 20
Participants | 0

3. Primary Outcome: Acute Procedural Success; Acute Vein Succes
Description: Demonstration of Acute Vein Success in all attempted PVs using the FARAPULSE Cardiac Ablation System Plus during the first ablation procedure (Index or Rescheduled Index Procedure)
Time Frame: Index Procedure
Measure: Number; unit: participants
Arm/Group | FARAPULSE™ Endocardial Cardiac Ablation
Number analyzed (Participants) | 20
participants | 20

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | FARAPULSE™ Endocardial Cardiac Ablation
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE™ Endocardial Cardiac Ablation (N=20)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE™ Endocardial Cardiac Ablation (N=20)
Hematoma (Vascular disorders) | 2 (2)
AV Fistula (Vascular disorders) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT05152966/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT05152966/SAP_001.pdf